## **Information for Patient**

## Prognostic Significance of Circulating Tumor DNA in Hodgkin Lymphoma

Dear patient,

We would like to invite you to participate in a laboratory research focused on Hodgkin lymphoma: its early diagnostics, and prediction of eventual tumor progression. This research is based on the analysis of circulating tumor DNA. Upon signing an informed consent, we would collect additional samples of your peripheral blood that will be taken together with regular blood tests related to your treatment in order to estimate the extent of the tumor and assess the prognosis.

Providing a sample of peripheral blood for molecular-genetic testing does not mean any additional medical risk, as it will be taken together with other routine diagnostic peripheral blood samples at the diagnosis and during the treatment.

Research of Hodgkin lymphoma is necessary for better understanding of its origin and behavior and critical for development of new therapeutic options in order to further improve its diagnostics and treatment.

Information obtained within this research will not be relevant for your current treatment, however, it could potentially improve early diagnostics or it could enhance development of new treatment options in patients with Hodgkin lymphoma in the future.

Providing a sample for molecular-genetic testing is entirely voluntary. If you do not wish to provide a sample, it would not negatively impact your medical care in any way. Analyses of samples and subsequent publications of results related to this research will be strictly anonymous and could not lead to individual patient identification.

Participation in this research does not entitle you to any compensatory payment.

All research data will be handled in accordance with regulations of the Czech Republic for protection of personal data and with corresponding EU legislation - the new General Data Protection Regulation (abbreviated GDPR) that was adopted and became effective on 25 May 2018. It replaces the Data Protection Directive (1995.

We ask you to give us a consent to process your selected disease related data. Only authorized staff involved in your regular health care would have an access to your medical records with your full identification data. This authorized staff has a duty of confidentiality based on the GDPR for personal data of patients.

Samples will be stored for research purposes during several years based on the advances of the research and related to research field. Samples will be labelled using codes, stored and processed anonymously in order to protect the personal data.

## **Informed Consent**

## Prognostic Significance of Circulating Tumor DNA in Hodgkin Lymphoma

I agree that the sample of peripheral blood can be used anonymously for research purposes.

This consent is given entirely voluntarily and I was informed that I can withdraw this consent at any time.

I acknowledge that no payment can be claimed by providing the sample of peripheral blood.

I agree that the results of blood samples analyses can be published in a scientific journal and can be potentially used for the development of new diagnostic procedures and for treatment follow-up. All results will be published anonymously in accordance with the relevant EU legislation- the General Data Protection Regulation that became effective on 25 May 2018.

I declare that I was informed about the research objective related to blood sample testing and that I received all additional information based on my questions.

| Name and Surname of the patient: |
|------------------------------------------------------------|
| Signature of the patient: |
| Place and date: |
| Name and Surname of the physician providing information: |
| Signature of treating the physician providing information: |
| Place and date: |
| Department: |